CLINICAL TRIAL: NCT02750462
Title: Immediate Unselected Coronary Angiography Versus Delayed Triage in Survivors of Out-of-hospital Cardiac Arrest Without ST-segment Elevation
Acronym: TOMAHAWK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Principal Investigator, Steffen Desch, Associate director, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOMAHAWK2.0
Record Dates: First submitted 2016-04-20; First posted 2016-04-25 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Out-of-hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate coronary angiography (Experimental): Immediate coronary angiography in survivors of out-of-hospital cardiac arrest without ST-segment elevation
  Interventions: Other: Immediate coronary angiography
- Delayed/selective coronary angiography (Active Comparator): Initial intensive care evaluation to further stratify the etiology of out-of-hospital cardiac arrest with delayed/selective coronary angiography if indicated
  Interventions: Other: Delayed/selective coronary angiography

INTERVENTIONS:
Other: Immediate coronary angiography — Immediate coronary angiography in survivors of out-of-hospital cardiac arrest without ST-segment elevation
  Arms: Immediate coronary angiography
Other: Delayed/selective coronary angiography — Initial intensive care evaluation to further stratify the etiology of out-of-hospital cardiac arrest with delayed/selective coronary angiography if indicated
  Arms: Delayed/selective coronary angiography

SUMMARY:
The aim of the trial is to compare immediate angiography in survivors of out of hospital cardiac arrest (OHCA) without ST-segment elevation versus delayed/selective catheterization with respect to 30 day mortality.

The TOMAHAWK trial is supported by the Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK).

DETAILED DESCRIPTION:
After inclusion and exclusion criteria have been checked patients will be randomized:

Group 1: Immediate angiography Patients randomized to group 1 will be transported to the catheterization laboratory as soon as possible after hospital admission for evaluation of coronary anatomy.

Group 2: Delayed/selective angiography Upon hospital admission, patients assigned to group 2 will first be transported to the ICU for further evaluation and stratification of OHCA etiology. Further triage will depend on the results of clinical examination and objective testing and will be left to the individual physician according to clinical judgment. Depending on clinical circumstances, further management may comprise medical therapy, laboratory testing, imaging such as echocardiography and/or computed tomography, hemodynamic or neurological monitoring, the initiation of therapeutic hypothermia or other measures of intensive care. If a high likelihood of an acute coronary trigger for OHCA persists (i.e. inconclusive results from clinical evaluation with ongoing suspicion of an acute coronary event, etc.), the treating physician may proceed to coronary angiography after a delay of 24h after the onset of cardiac arrest.

Vital status will be assessed at 30 days, 6 and 12 months after randomization by direct questioning if the patient is still hospitalized or structured telephone interview. Clinical events will be verified by original source data. At 6 and 12 months, quality of life will be assessed by the the Euroqol 5D questionnaire.

The TOMAHAWK trial is supported by the Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK).

ELIGIBILITY:
Inclusion Criteria:

* Documented resuscitated OHCA of possible cardiac origin and return of spontaneous circulation
* Age ≥30 years
* Informed consent

Exclusion Criteria:

* ST-segment elevation or new left bundle branch block
* No return of spontaneous circulation upon hospital admission
* Severe hemodynamic or electrical instability requiring immediate coronary angiography/intervention (delay clinically not acceptable)
* Obvious extra-cardiac etiology such as traumatic brain injury, primary metabolic or electrolyte disorders, intoxication, overt hemorrhage, respiratory failure due to known lung disease, suffocation, drowning
* In-hospital cardiac arrest
* Known or likely pregnancy
* Participation in another intervention study

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Universitäres Herzzentrum Lübeck, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rossberg M, Freund A, Thevathasan T, Skurk C, Koenig IR, Vens M, Grube H, Sandig F, Klinge K, Akin I, Fuernau G, Hassager C, Zeymer U, Preusch MR, Graf T, Jobs A, de Waha S, Thiele H, Poess J, Desch S. Quality of life after out-of-hospital cardiac arrest: a TOMAHAWK sub-study. Eur Heart J Acute Cardiovasc Care. 2025 Oct 7;14(9):511-519. doi: 10.1093/ehjacc/zuaf093. PMID 40557995
- [Derived] Spoormans EM, Thevathasan T, van Royen N, Zwinderman AH, Freund A, Thiele H, Ziesemer K, Desch S, Lemkes JS; COACT and TOMAHAWK Trials Investigators. One-Year Outcomes of Coronary Angiography After Out-of-Hospital Cardiac Arrest Without ST Elevation: An Individual Patient Data Meta-Analysis. JAMA Cardiol. 2025 Aug 1;10(8):779-786. doi: 10.1001/jamacardio.2025.1194. PMID 40434768
- [Derived] Desch S, Freund A, Akin I, Behnes M, Preusch MR, Zelniker TA, Skurk C, Landmesser U, Graf T, Eitel I, Fuernau G, Haake H, Nordbeck P, Hammer F, Felix SB, Hassager C, Kjaergaard J, Fichtlscherer S, Ledwoch J, Lenk K, Joner M, Steiner S, Liebetrau C, Voigt I, Zeymer U, Brand M, Schmitz R, Horstkotte J, Jacobshagen C, Poss J, Abdel-Wahab M, Lurz P, Jobs A, de Waha S, Olbrich D, Sandig F, Konig IR, Brett S, Vens M, Klinge K, Thiele H; TOMAHAWK Investigators. Coronary Angiography After Out-of-Hospital Cardiac Arrest Without ST-Segment Elevation: One-Year Outcomes of a Randomized Clinical Trial. JAMA Cardiol. 2023 Sep 1;8(9):827-834. doi: 10.1001/jamacardio.2023.2264. PMID 37556123
- [Derived] Desch S, Freund A, Akin I, Behnes M, Preusch MR, Zelniker TA, Skurk C, Landmesser U, Graf T, Eitel I, Fuernau G, Haake H, Nordbeck P, Hammer F, Felix SB, Hassager C, Engstrom T, Fichtlscherer S, Ledwoch J, Lenk K, Joner M, Steiner S, Liebetrau C, Voigt I, Zeymer U, Brand M, Schmitz R, Horstkotte J, Jacobshagen C, Poss J, Abdel-Wahab M, Lurz P, Jobs A, de Waha-Thiele S, Olbrich D, Sandig F, Konig IR, Brett S, Vens M, Klinge K, Thiele H; TOMAHAWK Investigators. Angiography after Out-of-Hospital Cardiac Arrest without ST-Segment Elevation. N Engl J Med. 2021 Dec 30;385(27):2544-2553. doi: 10.1056/NEJMoa2101909. Epub 2021 Aug 29. PMID 34459570
- [Derived] Desch S, Freund A, Graf T, Fichtlscherer S, Haake H, Preusch M, Hammer F, Akin I, Christ M, Liebetrau C, Skurk C, Steiner S, Voigt I, Schmitz R, Mudra H, Ledwoch J, Menck N, Horstkotte J, Pels K, Lahmann AL, Otto S, Lenk K, Ohlow MA, Hassager C, Nordbeck P, Zeymer U, Jobs A, de Waha-Thiele S, Olbrich D, Konig I, Klinge K, Thiele H. Immediate unselected coronary angiography versus delayed triage in survivors of out-of-hospital cardiac arrest without ST-segment elevation: Design and rationale of the TOMAHAWK trial. Am Heart J. 2019 Mar;209:20-28. doi: 10.1016/j.ahj.2018.12.005. Epub 2018 Dec 11. PMID 30639610